CLINICAL TRIAL: NCT04674163
Title: NEUROKINASE : Expression Profile of ERK5 and PKM2 Kinases in Neuroinflammatory Diseases.
Brief Title: Expression Profile of ERK5 and PKM2 Kinases in Neuroinflammatory Diseases.
Acronym: NEUROKINASE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no practitioner
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Collaborators: Immunologie et Neurogénétique Expérimentales et Moléculaires (INEM) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHRO-2018-07
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Sclerosis, Multiple; Guillain-Barre Syndrome; Inflammation
Keywords: ERK5 kinase; M2 Type Pyruvate Kinase; cytokines
MeSH Terms: conditions — Multiple Sclerosis; Guillain-Barre Syndrome; Inflammation | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with clinical signs that suggest Multiple Sclerosis (MS) or Guillain Barré Syndrome (GBS) (Experimental)
  Interventions: Biological: Blood sample and Cerebrospinal fluid (CSF) collection.

INTERVENTIONS:
Biological: Blood sample and Cerebrospinal fluid (CSF) collection. — An additional blood sample (25 ml) and a cerebrospinal fluid (CSF) sample (2 ml) will be taken.

SUMMARY:
Demyelinating diseases represent a broad spectrum of disorders and are induced by excessive inflammation most often triggered by an autoimmune mechanism. Some of these pathologies are chronic and affect the central nervous system such as multiple sclerosis (MS), others are monophasic and target the peripheral nervous system such as Guillain Barré syndrome (GBS).

In neuroinflammatory pathologies, the excessive response of the pro-inflammatory Th1 and Th17 lymphocyte lines and the insufficient response of regulatory T lymphocytes (Treg) cause excessive inflammation which is deleterious to the nervous tissue. The regulation of these signaling pathways involves key proteins such as kinases. Modulation of these kinases which could allow the development of new pharmacological targets for neuroinflammation.

Recent work (unpublished data) has shown an association between the expression of ERK5 and PMK2 kinases, and the clinical severity of experimental allergic encephalomyelitis, a mouse model that mimics multiple sclerosis.

In order to search for new biomarkers and improve our knowledge of the actors of the initial inflammatory phase of neuroinflammatory pathologies, we propose to study the differences in expression of ERK5 and PKM2 kinases in the blood and cerebral spinal fluid (CSF) of patients followed for relapsing-remitting MS and GBS by both RT-qPCR and protein quantification. We also want to study other biological parameters which include characterization of the pro / anti-inflammatory balance by cytokine assay and lymphocyte phenotyping, metabolome study, and mild form neurofilament (NfL) assay.

DETAILED DESCRIPTION:
The study of the expression of ERK5 and PKM2 kinases in patients followed for RR MS or GBS, at the beginning of the pathology, will be evaluate.

The usual diagnostic workup for MS and GBS will be performed in order to classify patients into 4 groups :

• Group 1 : control group. Patients that do not fulfill the criteria for MS or GBS and in whom no differential diagnosis was made.

Subgroups 1a and 1b will be formed by respective pairing with groups 2 and 3.

* Group 2 : patients with RR MS confirmed by Macdonald criteria (2017)
* Group 3 : patients with GBS confirmed by the association of the usual clinical and electrophysiological signs.
* Group 4 : patients in whom a differential diagnosis has been identified to explain the symptoms. These patients will be excluded from the analysis.

An additional blood sample (25 mL) and cerebrospinal fluid (CSF) sample (2mL) will be taken from all patients in order to study the laboratory parameters of this study. Peripheral blood mononuclear cells (PBMCs) and neutrophils will be isolated from the blood using a Percoll gradient. Group 4 samples will not be analyzed.

The analysis will focus on the comparison of laboratory parameters between group 2 and 3, between group 1a and 2, and between 1b and 3.

1. / Expression of ERK5 and PKM2 kinases

   The investigators wish to analyze the expression of ERK5 and PKM2 by RT-qPCR to investigate the transcriptome on RNA level and by Western Blot and ELISA to investigate the phosphorylated and total forms of the two kinases.

   RT-qPCR require RNA extraction, reverse transcription into cDNA and then amplification of the genes encoding ERK5 and PKM2 using specific primers designed beforehand. The results will be compared with those obtained with primers of the HPRT gene.
2. / Study of the balance between pro and anti-inflammatory action

   The investigators wish to characterize the balance of pro and anti-inflammatory activity by studying lymphocyte phenotyping and determining the level of cytokines.

   Lymphocyte phenotyping will be performed by flow cytometry from PBMCs. The populations studied will include the Th1, Th2, Th9, Th17, Th22, Treg and TFH populations.

   The panel of mainly inflammatory cytokines will be studied in plasma and in CSF by ELISA. The panel includes the following cytokines: IL17, TNF, IL6, Il 1β, IL 10, IL33, IL12, IL 23
3. / Metabolome analysis

   The databases on human metabolomes include more than 40,000 metabolites and allow the establishment of metabolic profiles in different pathological contexts by supervised and unsupervised statistical analysis techniques. Metabolome analyzes will be performed from plasma and CSF. These analyzes will be carried out by liquid chromatography coupled with mass spectrometry (LC-MS) by the Metabohub network (MetaboHUB-Clermont for plasma analyzes and MetaboHUB-Saclay for CSF analyzes).
4. / Measure of the neurofilament light chain (NfL)

There is growing interest in neurofilament's measure in the blood and in particular in the CSF. High levels of neurofilaments are evidence of neuronal loss, regardless of the initial mechanism. Neurofilament light chain (NfL) seems to be the most relevant form to measure axonal loss. In MS, increased NfL was observed during the first two months of acute relapse. Conversely, there are few data on the kinetics of NfL's levels in peripheral demyelinating diseases.

The investigators intend to study NfL levels in blood and CSF to determine if there is an increase in NfL levels in patients followed for GBS and to compare NfL levels of these patients (group 3) with patients followed for MS (group 2).

ELIGIBILITY:
Inclusion Criteria:

* Man and Woman
* 18 to 80 years old
* Clinical signs that suggest MS or GBS within a month of onset symptom

Exclusion Criteria:

* Patient treated with immunosuppressive therapy, immunomodulator, or corticosteroids in chronic treatment
* Patient treated with corticosteroids in the past month
* without social security
* HIV positive serology
* dementia
* pregnant or breastfeeding woman
* previous participation in the study
* under judicial protection
* non-cooperating patient

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Expression of genes encoding ERK5 and PKM2 kinases by RT-qPCR | Day 0
  The expression of ERK5 and PKM2 by RT-qPCR will be analyze to investigate the transcriptome on RNA level.
  RT-qPCR require RNA extraction, reverse transcription into cDNA and then amplification of the genes encoding ERK5 and PKM2 using specific primers designed beforehand. The results will be compared with those obtained with primers of the HPRT gene.
  These analyzes are carried out using lymphocytes and neutrophils isolated from the blood sample.

SECONDARY OUTCOMES:
Lymphocyte phenotyping | Day 0
  Lymphocyte phenotyping will be performed by flow cytometry from PBMCs. We will use antibodies against Th1, Th2, Th9, Th17, Th22, Treg and TFH populations.
Cytokine levels | Day 0
  A panel of cytokines, mainly pro-inflammatory, will be studied in plasma and in CSF by ELISA. The panel includes the following cytokines: IL17, TNF, IL6, Il 1β, IL 10, IL33, IL12, IL 23
Metabolome analysis | Day 0
  Metabolome analyzes will be performed from plasma and CSF. These analyzes will be carried out by liquid chromatography coupled with mass spectrometry (LC-MS) by the Metabohub network (MetaboHUB-Clermont for plasma analyzes and MetaboHUB-Saclay for CSF analyzes).
Measure of the neurofilament light chain (NfL) | Day 0
  NfL levels in blood and CSF will be studied to determine if there is an increase in NfL levels in patients followed for GBS and to compare the NfL levels of these patients with patients followed for MS.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal AUZOU, Dr, Principal Investigator — CHR Orléans

REFERENCES:
- [Background] Gaetani L, Salvadori N, Lisetti V, Eusebi P, Mancini A, Gentili L, Borrelli A, Portaccio E, Sarchielli P, Blennow K, Zetterberg H, Parnetti L, Calabresi P, Di Filippo M. Cerebrospinal fluid neurofilament light chain tracks cognitive impairment in multiple sclerosis. J Neurol. 2019 Sep;266(9):2157-2163. doi: 10.1007/s00415-019-09398-7. Epub 2019 May 25. PMID 31129709
- [Background] Kamil K, Yazid MD, Idrus RBH, Das S, Kumar J. Peripheral Demyelinating Diseases: From Biology to Translational Medicine. Front Neurol. 2019 Mar 19;10:87. doi: 10.3389/fneur.2019.00087. eCollection 2019. PMID 30941082
- [Background] Khalil M, Teunissen CE, Otto M, Piehl F, Sormani MP, Gattringer T, Barro C, Kappos L, Comabella M, Fazekas F, Petzold A, Blennow K, Zetterberg H, Kuhle J. Neurofilaments as biomarkers in neurological disorders. Nat Rev Neurol. 2018 Oct;14(10):577-589. doi: 10.1038/s41582-018-0058-z. PMID 30171200
- [Background] Kuhle J, Plattner K, Bestwick JP, Lindberg RL, Ramagopalan SV, Norgren N, Nissim A, Malaspina A, Leppert D, Giovannoni G, Kappos L. A comparative study of CSF neurofilament light and heavy chain protein in MS. Mult Scler. 2013 Oct;19(12):1597-603. doi: 10.1177/1352458513482374. Epub 2013 Mar 25. PMID 23529999
- [Background] Rostami A, Ciric B. Role of Th17 cells in the pathogenesis of CNS inflammatory demyelination. J Neurol Sci. 2013 Oct 15;333(1-2):76-87. doi: 10.1016/j.jns.2013.03.002. Epub 2013 Apr 8. PMID 23578791
- [Background] Thompson AJ, Banwell BL, Barkhof F, Carroll WM, Coetzee T, Comi G, Correale J, Fazekas F, Filippi M, Freedman MS, Fujihara K, Galetta SL, Hartung HP, Kappos L, Lublin FD, Marrie RA, Miller AE, Miller DH, Montalban X, Mowry EM, Sorensen PS, Tintore M, Traboulsee AL, Trojano M, Uitdehaag BMJ, Vukusic S, Waubant E, Weinshenker BG, Reingold SC, Cohen JA. Diagnosis of multiple sclerosis: 2017 revisions of the McDonald criteria. Lancet Neurol. 2018 Feb;17(2):162-173. doi: 10.1016/S1474-4422(17)30470-2. Epub 2017 Dec 21. PMID 29275977
- [Background] Venken K, Hellings N, Thewissen M, Somers V, Hensen K, Rummens JL, Medaer R, Hupperts R, Stinissen P. Compromised CD4+ CD25(high) regulatory T-cell function in patients with relapsing-remitting multiple sclerosis is correlated with a reduced frequency of FOXP3-positive cells and reduced FOXP3 expression at the single-cell level. Immunology. 2008 Jan;123(1):79-89. doi: 10.1111/j.1365-2567.2007.02690.x. Epub 2007 Sep 25. PMID 17897326
- [Background] Yuan A, Rao MV, Veeranna, Nixon RA. Neurofilaments and Neurofilament Proteins in Health and Disease. Cold Spring Harb Perspect Biol. 2017 Apr 3;9(4):a018309. doi: 10.1101/cshperspect.a018309. PMID 28373358